CLINICAL TRIAL: NCT03825900
Title: Transkranielle Gleichstromstimulation Und Die Interaktion Zwischen Chronischem Schmerz Und Der Intestinalen Epithelbarriere
Brief Title: Transcranial Direct Current Stimulation and the Interaction Between Chronic Pain and the Intestinal Epithelial Barrier in Patients With Chronic Inflammatory Bowel Diseases (IBD)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Magdalena S. Prüß née Volz, Principal Investigator, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA4/221/17
Record Dates: First submitted 2018-06-25; First posted 2019-02-01 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS (Active Comparator): Active transcranial direct current stimulation
  Interventions: Device: Sham OR active Transcranial direct current stimulation
- Sham tDCS (Sham Comparator): Sham transcranial direct current stimulation
  Interventions: Device: Sham OR active Transcranial direct current stimulation

INTERVENTIONS:
Device: Sham OR active Transcranial direct current stimulation — Sham OR active transcranial direct current stimulation over the motor cortex
  Other Names: Sham OR active tDCS

SUMMARY:
In the study the investigators aim to test whether transcranial direct current stimulation (tDCS) induced pain reduction is in association with functional changes in the brain measured with magnetic resonance imaging (MRI) and also with a change in permeability of the intestinal epithelial barrier in patients with chronic inflammatory bowel diseases (IBD)

Hypothesis: Transcranial direct current stimulation can reduce the perception of pain in patients with chronic inflammatory bowel diseases, which is in association with changes in the brain measured via MRI. Additionally, transcranial direct current stimulation and the induced pain reduction influence the permeability of the intestinal epithelial barrier

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease
* Chronic pain (more than 3 months)
* Pain (VAS > 3/10)

Exclusion Criteria:

* Contraindication to transcranial direct current stimulation
* Contraindications to functional magnetic resonance imaging (fMRI)
* Pregnancy
* Sever internal or psychiatric condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Functional changes in the brain measured with cerebral MRI | 6 weeks
  Exploratory analyses of resting-state fMRI
Structural changes in the brain measured with cerebral MRI | 6 weeks
  Exploratory analyses of MRI with respect to DTI (diffusions tensor imaging) and VBM (voxel based morphometry)
Functional and/or structural changes in the Intestinal Epithelial Barrier measured with endoscopy of the rectum with sample-taking | 6 weeks
Changes in pain measured with visual analogue scale | 6 weeks
  VAS , scale from 0-10
Changes in perception of pain measured with an algometer (pain pressure threshold) | 6 weeks
  continuous scale form 0 kg

SECONDARY OUTCOMES:
Changes in questionnaire "quality of life" | 6 weeks
  questionnaire "quality of life" analyses daily activities, scale running from 32 points (worse outcome) to 224 points (best outcome)
Changes in functional symptoms using IBS-SSS | 6 weeks
  IBS-SSS: irritable bowel syndrome - severity score system , questionnaire analyses functional symptoms, score running from 0 (best outcome) until 600 points (worst outcome)
Changes in activity indices using HWI questionnaire or SCCAI questionnaire | 6 weeks
  HWI: Harvey-Bradshaw-Index, SCCAI: Simple Clinical Colitis Activity Index, scale: points: 0-20 points (low points are best outcome, high points are worst outcome)
Changes in pain catastrophizing scale questionnaire | 6 weeks
  pain catastrophizing scale questionnaire analyses subjective catastrophizing due to pain, score running from 0-52 points (low points are best outcome, high points are worst outcome)
Changes in inflammation biomarker (blood - C-reactive protein) | 6 weeks
  unit: mg/dl
Changes in inflammation biomarker (stool - calprotectin) | 6 weeks
  Unit: mg/g

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena S Prüß-Volz, MD, Principal Investigator — Charite University
Locations (1):
- Charite University Medicine, Berlin, Germany